CLINICAL TRIAL: NCT01042184
Title: Phase IV Study Comparing the Duration of Sequential Therapy
Brief Title: Efficacy of 10-day and 14-day Sequential Therapy Versus Triple Therapy on the Eradication of Helicobacter Pylori
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200909054M; NTUH200909054M (Registry Identifier: NTUH); 200909054M
Record Dates: First submitted 2010-01-03; First posted 2010-01-05 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-06

CONDITIONS: H. Pylori Infection
Keywords: H. pylori infected patients without prior eradication therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): Group A: Sequential therapy for 14 days D1-D7: (lansoprazole 30mg + amoxicillin 1gm) bid D8-D14: (lansoprazole 30mg + clarithromycin 500mg + metronidazole 500mg) bid
  Interventions: Drug: Sequential therapy for 14 days
- Group B: Sequential therapy for 10 days (Experimental)
  Interventions: Drug: Sequential therapy for 10 days
- Group C: Triple therapy for 14 days (Active Comparator)
  Interventions: Drug: Triple therapy for 14 days

INTERVENTIONS:
Drug: Sequential therapy for 14 days — D1-D7: (lansoprazole 30mg + amoxicillin 1gm) bid D8-D14: (lansoprazole 30mg + clarithromycin 500mg + metronidazole 500mg) bi
  Arms: Group A
Drug: Sequential therapy for 10 days — D1-D5: (lansoprazole 30mg + amoxicillin 1gm) bid D6-D10: (lansoprazole 30mg+clarithromycin 500mg+metronidazole 500mg) bid
  Arms: Group B: Sequential therapy for 10 days
Drug: Triple therapy for 14 days — D1-D14: (lansoprazole 30mg + clarithromycin 500mg + amoxicillin 1gm) bid
  Arms: Group C: Triple therapy for 14 days

SUMMARY:
Background: Helicobacter pylori infection has been shown to be associated with the development of gastric cancer and peptic ulcer diseases. Eradication of H. pylori infection could reduce the occurence or recurrence of these diseases. However, the eradication rate of clarithromycin-based triple therapy has been declining in recent years, probably related to the increasing resistant rate to clarithromycin. It was estimated that 15-20% of patients would fail from first line standard eradication therapy and need second line rescue therapy. About 15-30% of patient would fail from second line therapy and need to be rescued with third line therapy. In recent years, the concept of sequential therapy has been advocated in the treatment of H. pylori infection. The regimen includes a PPI plus amoxicillin for five days, followed by a PPI plus clarithromycin and tinidazole for another five days. The eradication rate in the first line treatment of sequential therapy had been reported to be as high as 90%. More importantly, it has been demonstrated that the eradication rate among patients with clarithromycin-resistant strains could be as high as 89%. However, tinidazole is not available in many countries. Whether metronidazole would be an effective alternative to tinidazole in the sequential therapy remains unknown. Besides, whether extending the duration of sequential therapy from 10-day to 14-day would result in higher eradication rate also deserves further investigation. Furthermore, data on the efficacy of rescue regimens for patients who failed from first line sequential therapy are also lacking. The impact of clarithromycin, metronidazole resistance and CYP2C19 polymorphism on the sequential therapy containing metronidazole (rather than tinidazole) also has not been reported.

Aims: Therefore, we aim to assess

1. whether the substitution of metronidazole for tinidazole in the sequential therapy is also more effective than clarithromycin-based triple therapy
2. whether extending the duration of sequential therapy from 10-day to 14-day would achieve higher eradication rate
3. whether levofloxacin-based sequential therapy for 14-days is effective as second line rescue regimen for those who failed from first line sequential therapy
4. the impact of antibiotic resistance and CYP2C19 polymorphism on the eradication rate of sequential therapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients are aged greater than 20 years who have H. pylori infection without prior eradication therapy and are willing to receive the sequential therapy will be eligible for enrollment.

Exclusion Criteria:

1. children and teenagers aged less than 20 years,
2. history of gastrectomy,
3. gastric malignancy, including adenocarcinoma and lymphoma,
4. previous allergic reaction to antibiotics (amoxicillin, clarithromycin, levofloxacin, metronidazole) and prompt pump inhibitors (lansoprazole),
5. contraindication to treatment drugs,
6. pregnant or lactating women,
7. severe concurrent disease,
8. Patients who cannot give informed consent by himself or herself.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Eradication rate according to Intention to treat (ITT) and per-protocol (PP) analysis | 6 weeks after eradication therapy

SECONDARY OUTCOMES:
The impact of antibiotic resistance and CYP2C19 polymorphism on the eradication rate of sequential therapy | 6 weeks after eradication therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Ming Liou, M.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Liou JM, Chen CC, Chen MJ, Chen CC, Chang CY, Fang YJ, Lee JY, Hsu SJ, Luo JC, Chang WH, Hsu YC, Tseng CH, Tseng PH, Wang HP, Yang UC, Shun CT, Lin JT, Lee YC, Wu MS; Taiwan Helicobacter Consortium. Sequential versus triple therapy for the first-line treatment of Helicobacter pylori: a multicentre, open-label, randomised trial. Lancet. 2013 Jan 19;381(9862):205-13. doi: 10.1016/S0140-6736(12)61579-7. Epub 2012 Nov 16. PMID 23158886